CLINICAL TRIAL: NCT06229288
Title: Amoxicillin Alone Versus Amoxicillin/Clavulanate for Community-acquired Pneumonia in Patients Aged 65 Years or Older, and Hospitalized in a Non-intensive Care Unit Ward: a Non-inferiority Randomized Controlled Trial
Brief Title: Amoxicillin Alone Versus Amoxicillin/Clavulanate for Community-acquired Pneumonia in Patients Aged 65 Years or Older, and Hospitalized in a Non-intensive Care Unit Ward
Acronym: CAPTAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC20_0015
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Amoxicillin; Amoxicillin/clavulanate
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Amoxicillin; Drugs, Investigational; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: Drug study, multi-centre, Phase 3, Controlled , Randomized, Open, Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin (Experimental): Amoxicillin is an antibiotic treatment approved in France and in many countries.
  The investigational medicinal products (IMPs) are:
  - Amoxicillin capsules : Formulated as a 500 mg capsules for PO administration (commercially available). Description in IMP file.
  Amoxicillin capsules contain compendial excipients listed in the Summary Product Characteristics (SmPC), current version, and are kept in a cool dry place where the temperature stays at 15- 25°C.
  - Amoxicillin IV vials : Formulated as a 1000 mg vial for IV administration (commercially available). Description in IMP file.
  Amoxicillin IV vials contain compendial excipient listed in the Summary Product Characteristics (SmPC), current version, and are kept in a cool dry place where the temperature stays at 15-25°C.
  Interventions: Drug: Amoxicillin
- Amoxicillin/clavulanate (Active Comparator): Amoxicillin/clavulanate is recommended by French and European guidelines for the treatment of patients aged 65 years or older, and hospitalized in a non-ICU ward, as reported above.
  The active comparators (IMPs) are:
  - Amoxicillin/clavulanate tablets: Formulated as a tablet for PO administration (commercially available). Description in IMP file. Tablets contain 500 mg of amoxicillin trihydrate and 62.5 mg of clavulanate. Amoxicillin/clavulanate tablets contain compendial excipients listed in the Summary Product Characteristics (SmPC), current version, and are kept in a cool dry place where the temperature stays at 15-25°C.
  - Amoxicillin/clavulanate vials Vials contain 1000 mg of amoxicillin and 200 mg of clavulanate. Description in IMP file.
  Amoxicillin/clavulanate vials contain compendial excipients listed in the Summary Product Characteristics (SmPC), current version, and are kept in a cool dry place where the temperature stays at 15-25°C
  Interventions: Drug: Amoxicillin/clavulanate

INTERVENTIONS:
Drug: Amoxicillin — Participants will be randomized to IV/oral amoxicillin or IV/oral amoxicillin/clavulanate for 5 days. Both agents are approved for treatment of respiratory infections.
  Amoxicillin PO: The dose is two capsule of 500 mg every 8 hours (that is 3 times daily).
  Amoxicillin IV: The dose is 1 g every 8 hours (that is 3 times daily)
  Other Names: Experimental drug
  Arms: Amoxicillin
Drug: Amoxicillin/clavulanate — Participants will be randomized to IV/oral amoxicillin or IV/oral amoxicillin/clavulanate for 5 days. Both agents are approved for treatment of respiratory infections.
  Amoxicillin/clavulanate PO: The dose is two tablets of 500 mg/62.5 mg every 8 hours (that is 3 times daily, approved standard dose) Amoxicillin/clavulanate IV: The dose is 1 g/200 mg every 8 hours (that is 3 times daily, approved standard dose)
  Other Names: active comparator drug
  Arms: Amoxicillin/clavulanate

SUMMARY:
Reduce inappropriate antibiotic use is a priority of public health agencies. Community-acquired pneumonia (CAP) is one of the most important indications for antibiotic prescriptions.

In the majority of the studies of CAP, there is a large proportion of cases with no pathogen identified. Thus, the choice of the empirical antibiotic depends on the most likely pathogen, individual risk factors, comorbidities, and allergies.

Patients aged 65 years or older are often treated with amoxicillin/clavulanate or with another broad-spectrum antibiotic (third-generation cephalosporins, antipneumococcal fluoroquinolone). However, broad-spectrum antibiotic prescription in CAP is debated and concerns exist about side-effects and selective pressure for resistance. Due to lack of head-to-head antibiotic comparisons, a recent Cochrane review concluded that current evidence from Randomized Clinical Trials (RCTs) is insufficient to make evidence-based recommendations for the choice for antibiotic to be used, highlighting an important evidence gap.

DETAILED DESCRIPTION:
Thus, the goal of the proposed trial is to compare clinical efficacy and safety of two CAP antimicrobial treatments, amoxicillin and amoxicillin/clavulanate, in patients aged 65 years or older and hospitalized in a non-intensive care unit (ICU) ward. The CAPTAIN study will be a multi-center, randomized, open, non-inferiority trial comparing clinical efficacy at Day 30 among patients ≥65 years of age, and hospitalized in a non-ICU ward, treated with narrow-spectrum (amoxicillin) versus broad-spectrum (amoxicillin/clavulanate) antimicrobial therapy for CAP. This will be a pivotal clinical trial that will provide evidence to inform CAP treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 65 years or older with or without comorbidities defined by chronic diseases in immunocompetent patients,
2. Patient admitted to the hospital for a CAP defined by at least two clinical signs of pneumonia (cough, sputum production, dyspnea, tachypnea, or pleuritic pain, abnormal lung auscultatory sounds, fever (temperature > 38°C) or hypothermia (<36°C)), and had radiological evidence of a new infiltrate confirming pneumonia
3. Patient understanding oral and written French
4. Written informed consent obtained from patient prior to participation in the study (if the patient is unable to express in writing: consent by a trusted person).
5. Patients should be able to call and to answer to a phone call or to be with a relative who can help him to call or to answer questions notably raised by a medical staff belonging to the investigational site

Exclusion Criteria:

1. Signs of severe CAP (abscess, massive pleural effusion, serious chronic respiratory insufficiency, ICU admission)
2. Patient requiring ICU admission,
3. Estimated Glomerular Filtration Rate < 30 ml/min,
4. Known immunosuppression (asplenia, neutropenia, agammaglobulinemia, transplant, myeloma, lymphoma, known HIV and CD4<200/mm3),
5. Exacerbation of chronic obstructive pulmonary disease,
6. Life-threatening state expected to lead to possible imminent death,
7. Suspected atypical bacteria requiring combined antibiotics therapy,
8. Legionella suspected,
9. Subjects with clinical or epidemiological environment leading to suspect a healthcare associated pneumonia with antibiotic resistant pathogen (including long-term care facility)
10. Patient known to be colonized with Pseudomonas aeruginosa or Enterobacteriaceae in the respiratory tract,
11. Suspicion of aspiration pneumonia,
12. Administration of any antibiotic treatment for more than 24 hours before inclusion,
13. History of jaundice/hepatic impairment associated with amoxicillin/clavulanate acid,
14. History of bacterial pneumonia less than 1 month prior to study inclusion
15. History of hypersensitivity or allergy to beta-lactam or to any excipients included in study antibiotics,
16. Subject without health insurance,
17. Subject without home address or difficulty in terms of follow-up (vacation, job transfer, geographical distance, lack of motivation),
18. Patient under judicial protection,
19. Diagnosis confirmed of SAR-Cov2 infection (PCR Test, covid antigen rapid test, chest computed tomography (CT) scan),
20. Participation to another interventional study and having an exclusion period that is still in force during the screening phase or expected participation to another interventional study during participation to the CAPTAIN study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority | Day 30 after inclusion (=Day 1)
  To investigate non-inferiority in terms of clinical efficacy among patients aged 65 years or older, hospitalized in a non-ICU ward for a CAP, and treated with narrow-spectrum (amoxicillin) versus broad-spectrum (amoxicillin/clavulanate) antimicrobial therapy, at Day 30 since hospital admission. To answer this question, clinical success rate at Day 30 since admission, defined as survival after completion of antibiotic treatment course, resolution of signs and symptoms of the infection (cough, purulent sputum production, dyspnea, or pleuritic chest pain) present at baseline with no new symptoms or complications attributable to CAP and no need for further antibacterial therapy will be determined

SECONDARY OUTCOMES:
Rates of early clinical response | Day 3 after inclusion (=Day 1)
  Early clinical response will be defined as survival with improvement of one or more levels relative to baseline in two or more symptoms of CAP and no worsening of one or more levels in other symptoms of community-acquired bacterial pneumonia, without receipt of rescue antibacterial therapy
Clinical cure after the end of treatment | Within 30 days after inclusion (=Day 1) compared to baseline
  The proposed endpoint of clinical cure after the end of treatment is defined as resolution in relevant signs and symptoms reported at baseline, no worsening of symptoms, and no change in antimicrobial regimen
To investigate total duration of antibiotic treatment, i.e., the total number of days with antibiotics during the Day 30 follow-up after hospital admission | Day 30 after inclusion (=Day 1)
  Days taking antibiotics from the first dose until the interruption of any antibiotic treatment during hospitalization and at late follow-up at Day 30 after hospital admission (to identify the use of any other antibiotic after hospital discharge defined as no IV, regain of autonomy identical to baseline, good clinical response and favorable evolution following initiation of antibiotics, other criteria left at the discretion of the investigators according to centers' practices)
To investigate all-cause mortality at Day 30 after hospital admission | Day 30 after inclusion (=Day 1)
  All-cause mortality at Day 30 after hospital admission
To investigate the rate of polymerase chain reaction (PCR)-positive Clostridium difficile among patients with diarrhea | Within 30 days after inclusion (=Day 1)
  Number of positive polymerase chain reaction (PCR)-positive Clostridium difficile among patients with diarrhea
To investigate in-hospital mortality | Within 30 days after inclusion (=Day 1)
  Number of deaths during hospitalization
To investigate ICU transfer during the Day 30 follow-up | Day 30 after inclusion (=Day 1)
  Number of patients transferred to the ICU during the Day 30 follow-up
To investigate CAP recurrence and hospital readmissions up to day 30 from hospital admission | Day 30 after inclusion (=Day 1)
  Number of hospital readmissions and CAP recurrence up to day 30 from hospital admission
To investigate adverse events attributable to antibiotics up to day 30 from hospital admission | Day 30 after inclusion (=Day 1)
  Number of adverse events attributable to antibiotics and number of days with adverse events up to day 30 from hospital admission
To investigate compliance with the antibiotic treatment | Within 7 days after inclusion (=Day 1)
  Number of days of antibiotic treatment taken
To investigate length of hospital stay | Within 30 days after inclusion (=Day 1)
Analysis of sensitivity todiscordance | Within 30 days after inclusion (=Day 1)
  To investigate the agreement between the early clinical response endpoint and the investigator's clinical judgment: the agreement between early clinical response (main endpoint) and the investigator's clinical judgement (clinical success or clinical failure) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Frederic BALEN, Doctor, Principal Investigator — Toulouse UH; Guillaume MARTIN-BLONDEL, Doctor, Principal Investigator — Toulouse UH; Perrine DUMANOIR, Doctor, Principal Investigator — Grenoble Hospital; VIGLINO Damien, Doctor, Principal Investigator — Grenoble Hospital; Alexandrine VIDAL, Doctor, Principal Investigator — Perigueux Hospital; Delphine PLARD, Doctor, Principal Investigator — Angers UH; Rafaël MAHIEU, Doctor, Principal Investigator — Angers UH; Anne-Laure FERAL-PIERSSENS, Doctor, Principal Investigator — Avicenne AP-HP; Frederic MECHAI, Doctor, Principal Investigator — Avicenne AP-HP; Aurelie DAUMAS, Professor, Principal Investigator — Marseille Timone Hospital; Dominique MERRIEN, Doctor, Principal Investigator — CHD La Roche sur Yon; Sylvain LE GENTIL, Doctor, Principal Investigator — CHD La Roche sur Yon; Pierre BARSI, Doctor, Principal Investigator — Vannes Hospital Bretagne Atlantic; Rozenn LE BERRE, Doctor, Principal Investigator — Brest Hospital; Sylvain JAFFUEL, Doctor, Principal Investigator — Brest Hospital; Xavier DUBUCS, Doctor, Principal Investigator — Toulouse UH; Matthieu THIBAULT, Doctor, Principal Investigator — Saint-Nazaire Hospital; BOISSEAU Dorothée, Doctor, Principal Investigator — Saint-Nazaire Hospital
Locations (13):
- France (13):
  - CH Saint-Nazaire, Saint-Nazaire, France
  - Chu Angers, Angers
  - CHU Angers, Angers
  - CHU Avicenne AP-HP, Bobigny
  - CHRU Brest, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CHU Grenoble-Alpes, La Tronche
  - Assistance Publique Hopitaux De Marseille, Marseille
  - CHU de Nantes, Nantes
  - CH Perigueux, Périgueux
  - CHRU - TOULOUSE Hôpital Purpan, Toulouse
  - CHRU TOULOUSE - Hôpital Rangueuil, Toulouse
  - Centre Hospitalier Bretagne Atlantique, Vannes